CLINICAL TRIAL: NCT03623672
Title: North American Prodromal Synucleinopathy Consortium
Acronym: NAPS
Status: Enrolling by invitation | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Mayo Clinic (Other); University of Minnesota (Other); University of California, Los Angeles (Other); McGill University (Other); Emory University (Other); Massachusetts General Hospital (Other); National Institute on Aging (NIA) (NIH); Stanford University (Other); Portland VA Medical Center (U.S. Federal Agency); Banner Health (Other)
Responsible Party: Sponsor
Other Study IDs: 201712025; R34AG056639 (NIH)
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: REM Sleep Behavior Disorder; Parkinson Disease; Lewy Body Disease; Dementia With Lewy Bodies; Multiple System Atrophy; REM Sleep Parasomnias
Keywords: sleep; REM; rapid eye movement; parkinson; lewy body disease; dementia with lewy bodies; Multiple System Atrophy; parasomnia; synuclein; synucleinopathy
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease; Lewy Body Disease; Multiple System Atrophy; REM Sleep Parasomnias; Parasomnias; Synucleinopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood (plasma, buffy coat, extracted DNA) and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will enroll participants with idiopathic rapid eye movement (REM) sleep behavior disorder (RBD), for the purpose of preparing for a clinical trial of neuroprotective treatments against synucleinopathies.

DETAILED DESCRIPTION:
REM sleep behavior disorder (RBD) is a rare disorder where people act out their dreams. People with RBD often, but not always, develop Parkinson's Disease, dementia with Lewy bodies, multiple system atrophy, or other neurodegenerative diseases of the synucleinopathy type. The North American Prodromal Synucleinopathy (NAPS) Consortium was formed with the purpose of enrolling participants with RBD, in anticipation of a future clinical trial of a neuroprotective treatment against synucleinopathies. The NAPS Consortium will collect standardized clinical assessments, biofluids, and other data in order to develop biomarkers for synucleinopathies in the prodromal (presymptomatic) stage as well as a trial-ready registry of participants. Participants procedures will include a ~2-hour clinical assessment (medical history and physical exam), questionnaires, blood draw, and (at select sites) optional lumbar puncture.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic REM sleep behavior disorder

Exclusion Criteria:

* REM sleep behavior disorder secondary to another cause (ex: narcolepsy, dementia, Parkinson's Disease, etc)
* Other neurological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic REM sleep behavior disorder, adults.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-08-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Prodromal Synucleinopathy Rating Scale | 2 years
  Rating scale combining neurocognitive battery, motor, autonomic, olfaction, color vision functions. Global score range 0-3, with higher score indicating greater symptoms of synucleinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Yo-El Ju, MD, Principal Investigator — Washington University School of Medicine; Bradley Boeve, MD, Principal Investigator — Mayo Clinic
Locations (10):
- United States (9):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Redwood City, California
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Portland VA Medical Center, Portland, Oregon
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
This project will develop a large database of potential neurocognitive and polysomnographic biomarkers in rapid eye movement sleep behavior disorder (RBD), as well as a biobank of blood, DNA, and cerebrospinal fluid from individuals with RBD. Since individuals with RBD frequently develop synucleinopathies including Parkinson Disease, Dementia with Lewy Bodies (DLB), and Multiple System Atrophy, we anticipate that the data and samples we collect will be valuable for investigators interested in synucleinopathies, other dementias such as Alzheimer's Disease (AD), and sleep disorders. The neurocognitive battery will contain all components of the Uniform Dataset version 3 (UDS 3) with the additional DLB module, to harmonize with research efforts in AD and DLB. Biofluid samples will be banked at the National Cell Repository for Alzheimer's Disease (NCRAD) to facilitate distribution to other investigators.
Supporting Information: Study Protocol
Time Frame: Data will be made available after primary analyses planned by NAPS investigators in 2020. Data will be available indefinitely.
Access Criteria: IPD and sample requests will be determined by a Steering Committee
URL: http://naps-rbd.org

REFERENCES:
- [Derived] Postuma R, Vorasoot N, St Louis EK, Pelletier A, Lim MM, Elliott J, Gagnon JF, Gan-Or Z, Forsberg LK, Fields JA, Ross OA, Singer W, Huddleston DE, Bliwise DL, Avidan AY, Howell M, Schenck CH, McLeland J, Davis AA, Criswell SR, Videnovic A, During EH, Miglis MG, Boeve BF, Ju YS, McKeon A; as the North American Prodromal Synucleinopathy (NAPS) Consortium. IGLON5 Frequency in Idiopathic REM Sleep Behavior Disorder: A Multicenter Study. Neurol Neuroimmunol Neuroinflamm. 2024 Nov;11(6):e200311. doi: 10.1212/NXI.0000000000200311. Epub 2024 Sep 13. PMID 39270144
- [Derived] Elliott JE, Bryant-Ekstrand MD, Keil AT, Ligman BR, Lim MM, Zitser J, During EH, Gagnon JF, St Louis EK, Fields JA, Huddleston DE, Bliwise DL, Avidan AY, Schenck CH, McLeland J, Criswell SR, Davis AA, Videnovic A, Lee-Iannotti JK, Postuma R, Boeve BF, Ju YS, Miglis MG; for North American Prodromal Synucleinopathy (NAPS) Consortium. Frequency of Orthostatic Hypotension in Isolated REM Sleep Behavior Disorder. Neurology. 2023 Dec 12;101(24):e2545-e2559. doi: 10.1212/WNL.0000000000207883. Epub 2023 Oct 19. PMID 37857496